CLINICAL TRIAL: NCT02310672
Title: A Prospective, Multicenter, Single-arm, Open-label, Phase 4 Study to Evaluate the Effects of Macitentan on Right vEntricular Remodeling in Pulmonary ArterIal hypeRtension Assessed by Cardiac Magnetic Resonance Imaging
Brief Title: REPAIR: Right vEntricular Remodeling in Pulmonary ArterIal hypeRtension
Acronym: REPAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-403
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): All patients take open-label macitentan 10mg o.d.
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — All patients take open-label macitentan 10mg o.d.
  Other Names: ACT-064992

SUMMARY:
The study evaluates the effect of macitentan on right ventricular and hemodynamic properties in patients with symptomatic pulmonary arterial hypertension. Patients are treated with macitentan for 1 year. Patients undergo right heart catheterization (RHC) at baseline and Week 26. They also undergo cardiac magnetic resonance imaging (MRI) at baseline, Week 26 and Week 52. Safety is monitored throughout the study. The study has three stub-studies. Each patient can participate in no sub-study or in one sub-study. The sub-studies are: (1) metabolism sub-study (with PET-MR scans); (2) biopsy sub-study (biopsies taken during the RHC); (3) Echo sub-study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure
2. Symptomatic pulmonary arterial hypertension (PAH)
3. World Health Organization (WHO) Functional Class (FC) I to III
4. PAH etiology belonging to one of the following groups according to Nice classification:

   * Idiopathic PAH
   * Heritable PAH
   * Drug- and toxin-induced PAH
   * PAH associated with congenital heart diseases: only simple (atrial septal defect, ventricular septal defect, patent ductus arteriosus) congenital systemic to pulmonary shunts at least 2 year post surgical repair
5. Hemodynamic diagnosis of PAH confirmed by right heart catheterization (RHC) during screening showing:

   • mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg and
   * PCWP (pulmonary capillary wedge pressure) or left ventricular end diastolic pressure (LVEDP) ≤ 12 mmHg and pulmonary vascular resistance (PVR) ≥ 4 Wood Units (WU) (320 dyn.sec.cm-5) or
   * 12 mmHg ≤ PCWP or LVEDP ≤ 15 mmHg and PVR ≥ 6WU (480 dyn.sec.cm-5)
6. 6-minute walk distance (6MWD) ≥ 150 m during screening
7. For patients treated with oral diuretics, treatment dose must have been stable at least 1 month prior to RHC during the screening period
8. For patients treated with phosphodiesterase type-5 (PDE-5) inhibitors, treatment dose must have been stable at least 3 months prior to RHC during the screening period
9. For patients treated with beta blockers, treatment dose must have been stable at least 1 month prior to the RHC during the screening period
10. Men or women ≥18 and < 65 years
11. Women of childbearing potential (defined in protocol) must:

    * Have a negative serum pregnancy test during screening and a negative urine pregnancy test on Day 1, and
    * Agree to use reliable methods of contraception (defined in protocol) from screening up to 30 days after study treatment discontinuation, and
    * Agree to perform monthly pregnancy tests up to 30 days after study treatment discontinuation

Exclusion Criteria:

1. Body weight < 40 kg
2. Body mass index (BMI) > 35kg/m2. For patients with 30kg/m2 < BMI < 35kg/m2, an eligibility form will be submitted to a Steering Committee member who will reserve the right to exclude the patient.
3. Pregnancy, breastfeeding or intention to become pregnant during the study
4. Recently started (< 8 weeks prior to informed consent signature) or planned cardio-pulmonary rehabilitation program
5. Known concomitant life-threatening disease with a life expectancy < 12 months
6. Any condition likely to affect protocol or treatment compliance
7. Hospitalization for PAH within 3 months prior to informed consent signature
8. Left atrial volume indexed for body surface area ≥ 43mL/m2 by echocardiography or cardiac MRI
9. Valvular disease grade 2 or higher
10. History of pulmonary embolism or deep vein thrombosis
11. Documented moderate to severe chronic obstructive pulmonary disease
12. Documented moderate to severe restrictive lung disease
13. Historical evidence of significant coronary artery disease established by:

    * History of myocardial infarction or
    * More than 50% stenosis in a coronary artery (by percutaneous coronary intervention or angiography) or
    * Elevation of the ST segment on electrocardiogram or
    * History of coronary artery bypass grafting or
    * Stable angina
14. Diabetes mellitus
15. Moderate to severe renal insufficiency (calculated creatinine clearance < 60 mL/min/1.73 m2)
16. Cancer
17. Systolic blood pressure < 90 mmHg
18. Severe hepatic impairment (with or without cirrhosis) according to National Cancer Institute organ dysfunction working group criteria, defined as total bilirubin > 3 × upper limit of the normal range (ULN) accompanied by an aspartate aminotransferase (AST) elevation > ULN at Screening.
19. Hemoglobin < 100g/L
20. AST and/or alanine aminotransferase (ALT) > 3× ULN
21. Need for dialysis
22. Responders to acute vasoreactivity test based on medical history
23. Prior use of endothelin receptor antagonists (ERAs), stimulators of soluble guanylate cyclase or prostacyclin or prostacyclin analogues
24. Treatment with strong inducers of cytochrome P450 isozyme 3A4 (CYP3A4) within 4 weeks prior to study treatment initiation (e.g., carbamazepine, rifampicin, rifabutin, phenytoin and St. John's Wort)
25. Treatment with strong inhibitors of CYP3A4 within 4 weeks prior to study treatment initiation (e.g., ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, nefazodone, ritonavir, and saquinavir)
26. Treatment with another investigational drug (planned, or taken within the 3 months prior to study treatment initiation).
27. Hypersensitivity to any ERA or any excipients of the formulation of macitentan (lactose, magnesium stearate, microcrystalline cellulose, povidone, sodium starch glycolate, polyvinyl alcohol, polysorbate, titanium dioxide, talc, xanthan gum, and lecithin soya)
28. Claustrophobia
29. Permanent cardiac pacemaker, automatic internal cardioverter
30. Metallic implant (e.g., defibrillator, neurostimulator, hearing aid, permanent use of infusion device)
31. Atrial fibrillation, multiple premature ventricular or atrial contractions, or any other condition that would interfere with proper cardiac gating during MRI.
32. For patients enrolling in the metabolism sub-study only: glucose intolerance
33. For patients enrolling in the biopsy sub-study only: PAH etiology belonging to Nice classification 1.4.4: PAH associated with congenital heart diseases

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Perchenet, Study Director — Actelion
Locations (41):
- United States (8):
  - Massachussetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rudgers New Jersey Medical School, New Brunswick, New Jersey
  - Cornell University, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical, Dallas, Texas
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- The Prince Charles Hospital, Chermside, Queensland, Australia
- France (7):
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Michallon, La Tronche
  - "CHRU de Lille - Hôpital Albert Calmette ", Lille
  - Hopital de Brabois, Nancy
  - Hôpital Laennec, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital Européen Georges-Pompidou, Paris
- Germany (4):
  - Medizinische Klinik und Poliklinik II Universitätsklinik Bonn, Bonn
  - Universitätsklinikum Köln Herzzentrum / Klinik III für Innere Medizin, Cologne
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz Centrum für Thrombose und Hämostase, Mainz
- Hong Kong (3):
  - Grantham Hospital, Cardiac Medical Unit, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - United Christian Hospital, Hong Kong
- Israel (2):
  - Pulmonology institute, Soroka Medical Center, Beersheba
  - Shaare Zedek Medical Center, Jerusalem
- Italy (2):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Fondazione IRCCS Policlinico San Matteo Ambulatorio Scompenso Cardiaco e Trapianti, Pavia
- Malaysia (2):
  - Hospital Pulau Pinang, George Town
  - Institut Jantung Negara (National Heart Institute), Kuala Lumpur
- Netherlands (5):
  - VU University Medical Center (VUMC), Amsterdam
  - Maastricht UMC+, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Radboud UMC, Nijmegen
  - Erasmus University medical Center, Rotterdam
- Russia (2):
  - Russian Cardiology Scientific and Production Complex, Moscow
  - Almazov Federal North-West Medical Research Centre of Department of Health, Saint Petersburg
- Singapore (2):
  - National University Hospital - The Heart Institute - Cardiac Department, Singapore
  - National Heart Centre (NHC) Singapore, Singapore
- United Kingdom (3):
  - Golden Jubilee National Hospital, Glasgow
  - The Royal Free Hospital, London
  - "Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital", Sheffield

REFERENCES:
- [Derived] Kiely DG, Channick R, Flores D, Galie N, MacDonald G, Marcus JT, Mitchell L, Peacock A, Rosenkranz S, Tawakol A, Torbicki A, Vonk Noordegraaf A, Swift AJ. Comparison of cardiac magnetic resonance imaging, functional and haemodynamic variables in pulmonary arterial hypertension: insights from REPAIR. ERJ Open Res. 2024 Feb 12;10(1):00547-2023. doi: 10.1183/23120541.00547-2023. eCollection 2024 Jan. PMID 38348238
- [Derived] Torbicki A, Channick R, Galie N, Kiely DG, Moceri P, Peacock A, Swift AJ, Tawakol A, Vonk Noordegraaf A, Flores D, Martin N, Rosenkranz S. Effect of Macitentan in Pulmonary Arterial Hypertension and the Relationship Between Echocardiography and cMRI Variables: REPAIR Echocardiography Sub-study Results. Cardiol Ther. 2024 Mar;13(1):173-190. doi: 10.1007/s40119-023-00345-2. Epub 2024 Jan 28. PMID 38281309
- [Derived] Vonk Noordegraaf A, Channick R, Cottreel E, Kiely DG, Marcus JT, Martin N, Moiseeva O, Peacock A, Swift AJ, Tawakol A, Torbicki A, Rosenkranz S, Galie N. The REPAIR Study: Effects of Macitentan on RV Structure and Function in Pulmonary Arterial Hypertension. JACC Cardiovasc Imaging. 2022 Feb;15(2):240-253. doi: 10.1016/j.jcmg.2021.07.027. Epub 2021 Nov 17. PMID 34801462

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 112 participants were screened out of them 89 participants were enrolled in the study and of which 87 participants received study medication. Two participants who did not receive study treatment were wrongly classified as enrolled by the sites.
Groups:
- Macitentan 10 mg: Participants received macitentan 10 milligrams (mg) tablets once daily until the premature discontinuation of study drug or end of treatment (EOT) on the day of the last dose of study drug at Week 52.
Period: Overall Study
Arm/Group | Macitentan 10 mg
Started | 87
Completed | 72
Not Completed | 15
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Sponsor's decision | 12

BASELINE CHARACTERISTICS:
Population: Safety Set included all screened participants who received at least one dose of study drug.
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Asian | 26
  White | 46
  Other | 0
  Unknown or Not Reported | 14
Region of Enrollment [Count of Participants; unit: Participants]
  FRANCE | 14
  GERMANY | 12
  ISRAEL | 2
  ITALY | 3
  MALAYSIA | 8
  NETHERLANDS | 12
  RUSSIAN FEDERATION | 11
  SINGAPORE | 9
  UNITED KINGDOM | 3
  UNITED STATES | 6
  Hong Kong | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Right Ventricular Stroke Volume (RVSV) to Week 26
Description: Change from baseline in RVSV assessed by cardiac magnetic resonance imaging (MRI) from pulmonary artery flow was reported at Week 26. Primary analysis were based on interim results as pre-planned and the primary outcome measures data table reported is finalized as is.
Time Frame: Baseline and Week 26
Population: The Modified full analysis set (mFAS) included of all screened participants who received at least one dose of study drug and who had a baseline as well as a post-baseline measurement taken between 16 weeks and 30 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: milliliters (mL)
Groups:
- Macitanten 10 mg: Participants received macitentan 10 milligrams (mg) tablets once daily until the premature discontinuation of study drug or end of treatment (EOT) on the day of the last dose of study drug at Week 52.
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 42
milliliters (mL) | 15.17 (2.75)

2. Primary Outcome: Ratio of Week 26 to Baseline Pulmonary Vascular Resistance (PVR)
Description: Ratio of Week 26 to baseline PVR as assessed by RHC was reported. PVR represents the resistance against which the right ventricle needs to pump. PVR is determined by right heart catheterization (RHC). PVR was calculated as 80*(Mean pulmonary arterial pressure [mPAP] -[Pulmonary capillary wedge pressure {PCWP} or Left ventricular end diastolic pressure {LVEDP} if PCWP not available/cardiac output [CO]). Primary analysis were based on interim results as pre-planned and the primary outcome measures data table reported is finalized as is.
Time Frame: Baseline and Week 26
Population: mFAS included of all screened participants who received at least one dose of study drug and who had a baseline as well as a post-baseline measurement taken between 16 weeks and 30 weeks of treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 42
Ratio | 0.63 (0.11)

3. Secondary Outcome: Change From Baseline in Right Ventricular End Diastolic Volume (RVEDV) to Week 26
Description: Change from baseline to Week 26 in RVEDV assessed by cardiac MRI was reported.
Time Frame: Baseline to Week 26
Population: Safety set included all screened participants who received at least one dose of study drug. Here 'N' (number of participants analyzed) signifies the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 78
mL | -6.22 [-12.50 to 0.07]

4. Secondary Outcome: Change From Baseline in Right Ventricular End Systolic Volume (RVESV) to Week 26
Description: Change from baseline to Week 26 in RVESV assessed by cardiac MRI was reported.
Time Frame: Baseline to Week 26
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 78
mL | -16.39 [-20.56 to -12.21]

5. Secondary Outcome: Change From Baseline in Right Ventricular Ejection Fraction (RVEF) to Week 26 (% Blood Volume)
Description: Change from baseline to Week 26 in RVEF based on pulmonary artery flow assessed by cardiac MRI was reported.
Time Frame: Baseline to Week 26
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of blood volume
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 72
Percentage of blood volume | 10.14 [7.46 to 12.83]

6. Secondary Outcome: Change From Baseline in Right Ventricle (RV) Mass to Week 26
Description: Change from baseline to Week 26 in RV mass assessed by cardiac MRI was reported.
Time Frame: Baseline to Week 26
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Grams
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 78
Grams | -10.10 [-13.81 to -6.39]

7. Secondary Outcome: Change From Baseline in Six-minutes Walk Distance (6MWD) to Week 26
Description: 6MWD is a non-encouraged test performed in a 30 meter (m) long flat corridor, where the participant is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. This test is used to assess exercise capacity. The test was performed about 30 minutes after study drug administration. Any increase in the walk distance was considered improvement from baseline.
Time Frame: Baseline to Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 83
Meters | 38.85 (7.37)

8. Secondary Outcome: Change From Baseline in World Health Organization Functional Class (WHO FC) to Week 26
Description: WHO FC is a classification which reflects disease severity based on symptoms. WHO Functional Classification of pulmonary hypertension comprises of Class I (participants with pulmonary hypertension but without resulting limitation of physical activity), II (participants with pulmonary hypertension resulting in slight limitation of physical activity), III (participants with pulmonary hypertension resulting in marked limitation of physical activity) and IV (participants with pulmonary hypertension with inability to carry out any physical activity without symptoms). Changes from baseline to Week 26 included: improvement (change from a higher to a lower FC), worsening (change from a lower to a higher FC) or unchanged/stable (same FC at baseline and at the post-baseline time point).
Time Frame: Baseline to Week 26
Population: Safety Set included all screened participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitanten 10 mg
Number analyzed (Participants) | 87
Participants
  Missing WHO FC | 5
  Worsened WHO FC | 1
  Unchanged WHO FC | 35
  Improved WHO FC | 46

ADVERSE EVENTS:
Time Frame: Up to 420 Days
Description: Safety Set included all screened participants who received at least one dose of study drug.
Arm/Group | Macitentan 10 mg
All-Cause Mortality (participants affected / at risk) | 1/87
Serious Adverse Events (participants affected / at risk) | 15/87
Other Adverse Events (participants affected / at risk) | 57/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=87)
Anaemia (Blood and lymphatic system disorders) | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 2
Angina Pectoris (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 1
Ventricular Hypokinesia (Cardiac disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Therapeutic Response Decreased (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Cholangitis Infective (Infections and infestations) | 1
Cytomegalovirus Infection (Infections and infestations) | 1
Escherichia Bacteraemia (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Pelvic Haemorrhage (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=87)
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 6
Oedema Peripheral (General disorders) | 19
Pyrexia (General disorders) | 7
Nasopharyngitis (Infections and infestations) | 6
Upper Respiratory Tract Infection (Infections and infestations) | 10
Haemoglobin Decreased (Investigations) | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 8
Flushing (Vascular disorders) | 5

LIMITATIONS AND CAVEATS:
Due to the open-label non-comparative design of study, it cannot be excluded that 6MWD and WHO FC could have been influenced by participants' knowledge that they did receive an active treatment whose efficacy had already been demonstrated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT02310672/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT02310672/SAP_001.pdf